CLINICAL TRIAL: NCT06572358
Title: A Prospective, Open-label, Single-arm, Proof of Science, Clinical Safety and Efficacy Study of MetProUltima in Healthy Adult Human Subjects Having Symptoms of Gut Dysbiosis (Heart Burn, Bloating, Constipation, and Gut Immunity).
Brief Title: A Clinical Study to Assess the Safety and Effectiveness of Test Product in Healthy Adult Human Subjects Having Symptoms of Gut Dysbiosis (Heart Burn, Bloating, Constipation and Gut Immunity).
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NovoBliss Research Pvt Ltd (Other)
Collaborators: Meteoric Biopharmaceuticals Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NB240019-MB
Record Dates: First submitted 2024-08-11; First posted 2024-08-27 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Gut Dysbiosis

STUDY DESIGN:
Intervention Model Description: Prospective, Open-label, Single-arm, Proof of science
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MetProUltima (Experimental): Test product Name: MetProUltima Marketed By| Manufactured By: Meteoric Biopharmaceuticals Private Limited Mode of Usage: Take one capsule after each meal, twice daily. Frequency: Twice a Day Route of Administration: Oral
  Interventions: Other: MetProUltima

INTERVENTIONS:
Other: MetProUltima — Test product Name: MetProUltima Marketed By| Manufactured By: Meteoric Biopharmaceuticals Private Limited Mode of Usage: Take one capsule after each meal, twice daily. Frequency: Twice a Day Route of Administration: Oral

SUMMARY:
This is prospective, open-label, single-arm, proof of science, clinical safety and efficacy study of MetProUltima in healthy adult human subjects having symptoms of Gut Dysbiosis (heart burn, bloating, constipation).

DETAILED DESCRIPTION:
A total of up to 14 subjects will be enrolled to get 12 evaluable subjects complete the study.

The potential subjects will be screened as per the inclusion & exclusion criteria only after obtaining written informed consent from the subjects. Subjects having symptoms of gut dysbiosis like burning sensation, bloating nausea and altered bowel habit, digestion issues, aching joints and high tendency of falling sick, chronic fatigue, constipation, diarrhoea will be enrolled in the study. The subjects will be instructed to visit the facility as per the below visits.

Visit 01 (Day -01): Screening, Blood Sample Collection Visit 02 (Day 01): Enrolment, Faecal Sample Collection, Test Product Dispensing Visit 03 (Day 45 ±2 Days): Treatment usage period, Evaluations Visit 04 (Day 90 ±2 Days): Treatment usage period, Evaluations and End of study.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 to 65 years (both inclusive) at the time of consent.
2. Sex: Healthy males and healthy non-pregnant/non-lactating females.
3. Females of childbearing potential must have a self-reported negative pregnancy test.
4. Subject should have refrigerator at their home for storage of test product.
5. Subjects having history of falling sick frequently in two months.
6. Subjects having gut dysbiosis with either of these three symptoms which includes burning sensation, bloating, nausea, altered bowel habit, digestion issues, aching joints and high tendency of falling sick, chronic fatigue, constipation, diarrhoea etc.
7. If the subject is of childbearing potential, is practicing and agrees to maintain an established method of birth control (IUD, hormonal implant device/injection, regular use of birth control pills or patch, diaphragm, condoms with spermicide or sponge with spermicidal jelly, cream or foam, partner vasectomy or abstinence).
8. Subjects are willing to give written informed consent and are willing to come for regular follow-up.
9. Subjects who commit not to use other probiotics, symbiotic, prebiotics, medicated treatments or food having high probiotics other than the test product for the entire duration of the study.
10. Subject who has not participated in a similar investigation in the past three months.
11. Willing to use test product throughout the study period.

Exclusion Criteria:

1. Subject with suspected or proved organic causes of constipation, such as Hirschsprung's disease, hypothyroidism, or structural anomalies of the anal canal.
2. Subject with present condition of allergic response to any probiotic product.
3. Subjects under chronic medication (e.g. aspirin-based products, anti-inflammatories, anti-histamines, corticotherapy etc.) that might influence the outcome of the study.
4. Subjects with any major diseases of the cardiovascular, renal, hepatic, gastrointestinal, pulmonary or endocrine systems.
5. History of alcohol or drug addiction.
6. Subjects with a history of major gastrointestinal complications (i.e. Crohn's disease, ulcer, cancer, ulcerative colitis).
7. Subjects who have self-reported immuno-compromised (HIV positive, on anti-rejection medication, rheumatoid arthritis).
8. Pregnant or breastfeeding or planning to become pregnant during the study period.
9. Subjects participating in other similar product or therapeutic trials within the last four weeks.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2024-10-22 (Actual); Primary Completion 2025-02-07 (Actual); Study Completion 2025-02-07 (Actual)

PRIMARY OUTCOMES:
Changes in stool consistency based on the Bristol Stool Criteria | Baseline before usage of the test product on Day 01, and after usage of the test product on Day 45 and on Day 90
  To evaluate the effectiveness of the test product in terms of change in stool based on the Bristol Stool Criteria categorizes stools into one of seven stool types ranging from type 1 (hard lumps) to type 7 (watery diarrhoea).
Change in faecal microbiota using 16s Metagenome sequencing | Baseline at Day 1, and on Day 90.
  To evaluate the effectiveness of test product in terms of change in faecal microbiota using 16s Metagenome sequencing
Abbreviated physical examinations in terms of frequency of sensation of defecation | Baseline Day 1, Day 45 and on Day 90
  To evaluate the effectiveness of the test product by performing abbreviated physical examinations in terms of frequency of sensation of defecation according to a 5-point Likert scale, with a score ranging from 0 (no symptoms) to 20 (very severe symptoms
Abbreviated physical examinations in terms of bloating | Baseline Day 1, Day 45 and on Day 90
  To evaluate the effectiveness of the test product by performing abbreviated physical examinations in terms of bloating in which scoring done as less than 1 week=1, less than1 month=2, less than 2 months=3 and more than 2 months=4
Abbreviated physical examinations in terms of nausea | Baseline Day 1, Day 45 and on Day 90
  To evaluate the effectiveness of the test product by performing abbreviated physical examinations in terms of nausea where scoring determined no nausea=0, mild nausea=1-2, moderate nausea 3-6, and severe nausea7-9
Abbreviated physical examinations in terms of altered bowel habit. | Baseline Day 1, Day 45 and on Day 90
  To evaluate the effectiveness of the test product by performing abbreviated physical examinations in terms of altered bowel habit in which scoring done as less than 1 week=1, less than1 month=2, less than 2 months=3 and more than 2 months=4
Abbreviated physical examinations in terms of digestion issues | Baseline Day 1, Day 45 and on Day 90
  To evaluate the effectiveness of the test product by performing abbreviated physical examinations in terms of digestion issues in which scoring done on yes or no
Abbreviated physical examinations in terms of aching joints | Baseline Day 1, Day 45 and on Day 90
  To evaluate the effectiveness of the test product by performing abbreviated physical examinations in terms of aching joints in which scoring done as less than 1 week=1, less than1 month=2, less than 2 months=3 and more than 2 months=4
Abbreviated physical examinations in terms of chronic fatigue | Baseline Day 1, Day 45 and on Day 90
  To evaluate the effectiveness of the test product by performing abbreviated physical examinations in terms of chronic fatigue in which scoring done as less than 1 week=1, less than1 month=2, less than 6 months=3 and more than 6 months=4
Abbreviated physical examinations in terms of constipation for Frequency of bowel movements | Baseline Day 1, Day 45 and on Day 90
  To evaluate the effectiveness of the test product by performing abbreviated physical examinations in terms of constipation for Frequency of bowel movements in which scoring done 1-2 times per 1-2 days=1 and less than once per month=4
Abbreviated physical examinations in terms of constipation for Completeness: feeling incomplete evacuation | Baseline Day 1, Day 45 and on Day 90
  To evaluate the effectiveness of the test product by performing abbreviated physical examinations in terms of constipation for Completeness: feeling incomplete evacuation in which scoring done never=0 and always=4
Abbreviated physical examinations in terms of constipation for Time: minutes in lavatory per attempt | Baseline Day 1, Day 45 and on Day 90
  To evaluate the effectiveness of the test product by performing abbreviated physical examinations in terms of constipation for Time: minutes in lavatory per attempt in which scoring done Less than 5=0 and More than 30=4
Abbreviated physical examinations in terms of constipation for Failure: unsuccessful attempts for evacuation per 24 hours | Baseline Day 1, Day 45 and on Day 90
  To evaluate the effectiveness of the test product by performing abbreviated physical examinations in terms of constipation for Failure: unsuccessful attempts for evacuation per 24 hours in which scoring done never=0 and More than 9 =4
Abbreviated physical examinations in terms of constipation for Difficulty: painful evacuation effort | Baseline Day 1, Day 45 and on Day 90
  To evaluate the effectiveness of the test product by performing abbreviated physical examinations in terms of constipation for Difficulty: painful evacuation effort in which scoring done never=0 and always =4
Abbreviated physical examinations in terms of constipation for Pain: abdominal pain | Baseline Day 1, Day 45 and on Day 90
  To evaluate the effectiveness of the test product by performing abbreviated physical examinations in terms of constipation for Pain: abdominal pain in which scoring done never=0 and always =4
Abbreviated physical examinations in terms of constipation for Assistance: type of assistance | Baseline Day 1, Day 45 and on Day 90
  To evaluate the effectiveness of the test product by performing abbreviated physical examinations in terms of constipation for Assistance: type of assistance in which scoring done without assistance=0 and Digital assistance or enema =2
Abbreviated physical examinations in terms of constipation for History: duration of constipation (years) | Baseline Day 1, Day 45 and on Day 90
  To evaluate the effectiveness of the test product by performing abbreviated physical examinations in terms of constipation for History: duration of constipation (years) in which scoring done 0=0 and more than 20 =4
Abbreviated physical examinations in terms of diarrhoea | Baseline Day 1, Day 45 and on Day 90
  To evaluate the effectiveness of the test product by performing abbreviated physical examinations in terms of diarrhoeawhere score, severe diarrhea - having more than 10 loose, watery stools in a single day (24 hours). Moderate diarrhea -having more than a few but not more than 10 diarrhea stools in a day and Mild

SECONDARY OUTCOMES:
Effectiveness by biomarkers like CRP (C reactive protein). | baseline Day 01 and after usage of the test product on Day 90.
  To assess the effectiveness of the test product by Biomarkers like CRP(C reactive protein)
Effectiveness by biomarkers like IL-6 (Interleukin-6). | baseline Day 01 and after usage of the test product on Day 90.
  To assess the effectiveness of the test product by Biomarkers IL-6 (Interleukin-6)
Effectiveness of the test product in terms of subject perception questionnaire where scoring by licert scale where 1 = not at all and 5=Extremely | Baseline before usage of the test product on Day 01 and after usage of the test product, on Day 45 and on Day 90
  To assess the effectiveness of the test product in terms of subject perception questionnaire
change in lab parameters-Hemoglobin | Baseline on Day -01 and after usage of the test product on Day 90.
  To assess the effectiveness of the test product in terms of change in lab parameters Hemoglobin
change in lab parameters-Hematocrit | Baseline on Day -01 and after usage of the test product on Day 90.
  To assess the effectiveness of the test product in terms of change in lab parameters Hematocrit
change in lab parameters-RBC Counts (Red Blood Corpuscle) | Baseline on Day -01 and after usage of the test product on Day 90.
  To assess the effectiveness of the test product in terms of change in lab parameters RBC Counts (Red Blood Corpuscle)
change in lab parameters-MCV (Mean corpuscular volume) | Baseline on Day -01 and after usage of the test product on Day 90.
  To assess the effectiveness of the test product in terms of change in lab parameters MCV (Mean corpuscular volume)
change in lab parameters-MCH (mean corpuscular hemoglobin) | Baseline on Day -01 and after usage of the test product on Day 90.
  To assess the effectiveness of the test product in terms of change in lab parameters MCH (mean corpuscular hemoglobin)
change in lab parameters-MCHC (Mean corpuscular hemoglobin concentration) | Baseline on Day -01 and after usage of the test product on Day 90.
  To assess the effectiveness of the test product in terms of change in lab parameters MCHC (Mean corpuscular hemoglobin concentration)
change in lab parameters-RDW (Red cell distribution width) | Baseline on Day -01 and after usage of the test product on Day 90.
  To assess the effectiveness of the test product in terms of change in lab parameters RDW (Red cell distribution width)
change in lab parameters-WBC Counts (White blood cells) | Baseline on Day -01 and after usage of the test product on Day 90.
  To assess the effectiveness of the test product in terms of change in lab parameters WBC Counts (White blood cells)
change in lab parameters-Neutrophils | Baseline on Day -01 and after usage of the test product on Day 90.
  To assess the effectiveness of the test product in terms of change in lab parameters Neutrophils
change in lab parameters-Lymphocytes | Baseline on Day -01 and after usage of the test product on Day 90.
  To assess the effectiveness of the test product in terms of change in lab parameters Lymphocytes
change in lab parameters-Eosinophils | Baseline on Day -01 and after usage of the test product on Day 90.
  To assess the effectiveness of the test product in terms of change in lab parameters Eosinophils
change in lab parameters-Monocytes | Baseline on Day -01 and after usage of the test product on Day 90.
  To assess the effectiveness of the test product in terms of change in lab parameters Monocytes
change in lab parameters-Basophils | Baseline on Day -01 and after usage of the test product on Day 90.
  To assess the effectiveness of the test product in terms of change in lab parameters Basophils
change in lab parameters-RBC morphology | Baseline on Day -01 and after usage of the test product on Day 90.
  To assess the effectiveness of the test product in terms of change in lab parameters RBC morphology
change in lab parameters-Platelet Count | Baseline on Day -01 and after usage of the test product on Day 90.
  To assess the effectiveness of the test product in terms of change in lab parameters Platelet Count
change in lab parameters-Random Blood Sugar | Baseline on Day -01 and after usage of the test product on Day 90.
  To assess the effectiveness of the test product in terms of change in lab parameters Random Blood Sugar
change in lab parameters-Total Serum Cholesterol | Baseline on Day -01 and after usage of the test product on Day 90.
  To assess the effectiveness of the test product in terms of change in lab parameters Total Serum Cholesterol
change in lab parameters-Triglyceride | Baseline on Day -01 and after usage of the test product on Day 90.
  To assess the effectiveness of the test product in terms of change in lab parameters Triglyceride
change in lab parameters-HDL (High-density lipoprotein cholesterol) | Baseline on Day -01 and after usage of the test product on Day 90.
  To assess the effectiveness of the test product in terms of change in lab parameters HDL (High-density lipoprotein cholesterol)
change in lab parameters-LDL (Low-density lipoprotein) | Baseline on Day -01 and after usage of the test product on Day 90.
  To assess the effectiveness of the test product in terms of change in lab parameters LDL (Low-density lipoprotein)
change in lab parameters-Serum Creatinine | Baseline on Day -01 and after usage of the test product on Day 90.
  To assess the effectiveness of the test product in terms of change in lab parameters Serum Creatinine
change in Urine Routine and Microscopy -Color | Baseline on Day -01 and after usage of the test product on Day 90.
  To assess the effectiveness of the test product in terms of change in Urine Routine and Microscopy -Color
change in Urine Routine and Microscopy -Transparency | Baseline on Day -01 and after usage of the test product on Day 90.
  To assess the effectiveness of the test product in terms of change in Urine Routine and Microscopy -Transparency
change in Urine Routine and Microscopy -Specific Gravity | Baseline on Day -01 and after usage of the test product on Day 90.
  To assess the effectiveness of the test product in terms of change in Urine Routine and Microscopy -Specific Gravity
change in Urine Routine and Microscopy -pH | Baseline on Day -01 and after usage of the test product on Day 90.
  To assess the effectiveness of the test product in terms of change in Urine Routine and Microscopy -pH
change in Urine Routine and Microscopy -Albumin | Baseline on Day -01 and after usage of the test product on Day 90.
  To assess the effectiveness of the test product in terms of change in Urine Routine and Microscopy -Albumin
change in Urine Routine and Microscopy -Glucose | Baseline on Day -01 and after usage of the test product on Day 90.
  To assess the effectiveness of the test product in terms of change in Urine Routine and Microscopy -Glucose
change in Urine Routine and Microscopy -Bile Salts | Baseline on Day -01 and after usage of the test product on Day 90.
  To assess the effectiveness of the test product in terms of change in Urine Routine and Microscopy -Bile Salts
change in Urine Routine and Microscopy -Bile Pigments | Baseline on Day -01 and after usage of the test product on Day 90.
  To assess the effectiveness of the test product in terms of change in Urine Routine and Microscopy -Bile Pigments
change in Urine Routine and Microscopy -Bilirubin | Baseline on Day -01 and after usage of the test product on Day 90.
  To assess the effectiveness of the test product in terms of change in Urine Routine and Microscopy -Bilirubin
change in Urine Routine and Microscopy -Urobilinogen | Baseline on Day -01 and after usage of the test product on Day 90.
  To assess the effectiveness of the test product in terms of change in Urine Routine and Microscopy -Urobilinogen
change in Urine Routine and Microscopy -Ketone | Baseline on Day -01 and after usage of the test product on Day 90.
  To assess the effectiveness of the test product in terms of change in Urine Routine and Microscopy -Ketone
change in Urine Routine and Microscopy -Nitrite | Baseline on Day -01 and after usage of the test product on Day 90.
  To assess the effectiveness of the test product in terms of change in Urine Routine and Microscopy -Nitrite
change in Urine Routine and Microscopy -RBCs (Red Blood Corpuscle) | Baseline on Day -01 and after usage of the test product on Day 90.
  To assess the effectiveness of the test product in terms of change in Urine Routine and Microscopy -RBCs (Red Blood Corpuscle)
change in Urine Routine and Microscopy -Leucocyte | Baseline on Day -01 and after usage of the test product on Day 90.
  To assess the effectiveness of the test product in terms of change in Urine Routine and Microscopy -Leucocyte
change in Urine Routine and Microscopy -WBC (White blood cell) | Baseline on Day -01 and after usage of the test product on Day 90.
  To assess the effectiveness of the test product in terms of change in Urine Routine and Microscopy -WBC (White blood cell)
change in Urine Routine and Microscopy -Epithelial Cell | Baseline on Day -01 and after usage of the test product on Day 90.
  To assess the effectiveness of the test product in terms of change in Urine Routine and Microscopy -Epithelial Cell
change in Urine Routine and Microscopy -Casts | Baseline on Day -01 and after usage of the test product on Day 90.
  To assess the effectiveness of the test product in terms of change in Urine Routine and Microscopy -Casts
change in Urine Routine and Microscopy -Crystals | Baseline on Day -01 and after usage of the test product on Day 90.
  To assess the effectiveness of the test product in terms of change in Urine Routine and Microscopy -Crystals
Adverse events | Baseline Day 1, Day 45 and on Day 90
  Safety will be determined by treatment-emergent adverse events such as allergies, diarrhoea, bloating, nausea, headache assessed by the study investigator.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Nayan K Patel, Principal Investigator — NovoBliss Research Pvt Ltd
Locations (1):
- NovoBliss Research Pvt.Ltd, Ahmedabad, Gujarat, India

IPD SHARING:
Plan to Share IPD: No